CLINICAL TRIAL: NCT00849758
Title: Gene Polymorphisms and Gene Products as Biological Markers of Aging and Correlation With Clinical Geriatric Assessment, Tolerance of Chemotherapy and Outcome in Elderly Breast Cancer Patients.
Acronym: EBS
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Hans Wildiers, adjunct head of clinic, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S51518
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Breast Cancer; Elderly
Keywords: breast cancer; elderly; biomarker
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood is collected for DNA, RNA, serum plasma, and lymphocytes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: chemotherapy: elderly patients receiving 4x adjuvant taxotere cyclophosphamide adjuvant for breast cancer
- 2: adjuvant hormone therapy: 40 patients receiving adjuvant aromatase inhibitor without chemotherapy

SUMMARY:
The goal is to study the biology of aging in breast cancer patients, and to study the impact of chemotherapy on aging related blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 70 years or older
* Female
* Early breast cancer
* Candidate for systemic adjuvant therapy

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: 70+, female, M0, all breast tumor types allowed (main goal is effect of chemo on the patient; looking at ER pos only would lead to insufficient numbers).
  80 patients receiving adjuvant TC (taxotere cyclophosphamide 75/600) q3w, 4x Nadir systematically in first cycle (d10 and 15) to have idea on haematological toxicity grades III-IV.
  No primary prophylaxis at first cycle, but allowed for secondary prophylaxis (febrile neutropenia or prolonged neutropenia = 5d < 500 neutrophils).
  Herceptin preferably given in HER2 positive patients after chemo (HERA like) in order to have similar treatment; but the investigator can also give concomitantly with chemo.
  40 patients receiving 5y AI (control group).
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-05; Primary Completion 2012-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
the primary question is whether Chemotherapy affects biological aging markers, such as telomere length and immune status | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - Jules Bordet Institute, Brussels
  - University Hospitals Leuven, Leuven

REFERENCES:
- [Derived] Dalmasso B, Hatse S, Brouwers B, Laenen A, Berben L, Kenis C, Smeets A, Neven P, Schoffski P, Wildiers H. Age-related microRNAs in older breast cancer patients: biomarker potential and evolution during adjuvant chemotherapy. BMC Cancer. 2018 Oct 22;18(1):1014. doi: 10.1186/s12885-018-4920-6. PMID 30348127
- [Derived] Bailur JK, Pawelec G, Hatse S, Brouwers B, Smeets A, Neven P, Laenen A, Wildiers H, Shipp C. Immune profiles of elderly breast cancer patients are altered by chemotherapy and relate to clinical frailty. Breast Cancer Res. 2017 Feb 28;19(1):20. doi: 10.1186/s13058-017-0813-x. PMID 28241844